CLINICAL TRIAL: NCT04333069
Title: Outcome of Cataract Surgery in Patient With Uveitis
Brief Title: Outcome of Cataract Surgery With Uveitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Abdallah Abdal Razik Ahmed, Assistant lecturer at Ophthalmology departmentAssiut University Faculty of Medicine, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: cat in uveitic patients
Record Dates: First submitted 2020-03-28; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Cataract; Complicata
Keywords: uveitis
MeSH Terms: conditions — Cataract; Uveitis | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uncorrected and best corrected visual acuity (Other): Measuring of uncorrected and best corrected visual acuity after phaco emulsification and irrigation aspiration cataract surgery
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — cataract surgery in form of phaco emulsification or irrigation aspiration

SUMMARY:
Aim of the study is to evaluate outcome of cataract surgery in different types of uveitis as regarding best corrected visual acuity (BCVA) and rate of post operative complications.

DETAILED DESCRIPTION:
Cataract is the main cause of reversible blindness in patients with uveitis. Cataract occurs in up to 50% to 70% of patients with uveitis.

Preoperative complications, including anterior synechiae, posterior synechiae, and pupillary membrane formation, may increase surgical challenges. In addition, recurrent inflammation increases the incidence of postoperative complications and often affects the visual prognosis. In recent years, phacoemulsification with intra ocular lens (IOL)implantation has become the main surgical method for treating uveitis (complicated cataract), and the visual prognosis of patients who undergo this procedure is usually favorable.

Surgical treatment may be effective but is associated with higher rates of complication than in non uveitic eyes. Cystoid macular edema (CME) is the most common complication cataract surgery in the general population. Although, in most cases, the macular edema is self-limited, in rare cases it can lead to long-term visual deterioration that is difficult to treat.

Another common complication after cataract surgery is posterior capsule opacification (PCO) , leading to symptoms of glare or blurred vision, reduced visual acuity, or impaired posterior segment exam. Factors that are critical in the development of PCO include surgical technique, type of implanted intra ocular lens (IOL) either foldable hydrophilic acrylic, hydrophobic acrylic or silicone and postoperative control of uveitis

ELIGIBILITY:
Inclusion Criteria:

- Visually significant cataract ( means opacification of the crystalline lens adequate to interfere with vision)in patients with uveitis controlled for at least 1month.

Exclusion Criteria:

* Irreversible pathology affecting outcome e.g. macular scar ,optic atrophy, and retinal detachment.
* Patients with active uveitis (means inflammation inside the eye).
* Patients less than 16 years old.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-10 (Estimated); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
final postoperative uncorrected visual acuity (UCVA) | 1 week post operative
  post operative uncorrected visual acuity which mean visual acuity without spectacle correction
final postoperative uncorrected visual acuity (UCVA) | 1month post operative
  post operative uncorrected visual acuity which mean visual acuity without spectacle correction
final postoperative uncorrected visual acuity (UCVA) | 3months post operative
  post operative uncorrected visual acuity which mean visual acuity without spectacle correction
final postoperative uncorrected visual acuity (UCVA) | 6months post operative
  post operative uncorrected visual acuity which mean visual acuity without spectacle correction
Final post operative best corrected visual acuity (BCVA) | 1 week post operative
  Post operative visual acuity with spectacle correction
Final post operative best corrected visual acuity (BCVA) | 1month post operative
  Post operative visual acuity with spectacle correction
Final post operative best corrected visual acuity (BCVA) | 3months post operative
  Post operative visual acuity with spectacle correction
Final post operative best corrected visual acuity (BCVA) | 6months post operative
  Post operative visual acuity with spectacle correction

SECONDARY OUTCOMES:
incidence of postoperative complications | 6 months post operative
  cystoid macular edema which mean inflammation, swelling and collection of fluid inside macula) .
Reactivation of intraocular inflammation | 6 months post operative
  Appearance of inflammatory activity inside the eye after period of quiescence of at least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Khalaf Al Husseini, professor, Study Director — Assiut University; Wael Mohammed Ahmed Soliman, professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpentier SJ, Jung JL, Patnaik JL, Pecen PE, Palestine AG. A Cross-Sectional Online Survey Identifies Subspecialty Differences in the Management of Pediatric Cataracts Associated with Uveitis. Ophthalmol Ther. 2020 Jun;9(2):293-303. doi: 10.1007/s40123-020-00245-x. Epub 2020 Mar 10. PMID 32157612
- [Background] Chen JL, Bhat P, Lobo-Chan AM. Perioperative Management of Uveitic Cataracts. Adv Ophthalmol Optom. 2019 Aug;4:325-339. doi: 10.1016/j.yaoo.2019.04.014. Epub 2019 May 18. PMID 31788579
- [Background] Yangzes S, Seth NG, Singh R, Gupta PC, Jinagal J, Pandav SS, Gupta V, Gupta A, Ram J. Long-term outcomes of cataract surgery in children with uveitis. Indian J Ophthalmol. 2019 Apr;67(4):490-495. doi: 10.4103/ijo.IJO_846_18. PMID 30900580
- [Background] Jinagal J, Gupta G, Agarwal A, Aggarwal K, Akella M, Gupta V, Suri D, Gupta A, Singh S, Ram J. Safety and efficacy of dexamethasone implant along with phacoemulsification and intraocular lens implantation in children with juvenile idiopathic arthritis associated uveitis. Indian J Ophthalmol. 2019 Jan;67(1):69-74. doi: 10.4103/ijo.IJO_713_18. PMID 30574896
- [Background] El Gharbawy SA, Darwish EA, Abu Eleinen KG, Osman MH. Efficacy of addition of nepafenac 0.1% to steroid eye drops in prevention of post-phaco macular edema in high-risk eyes. Eur J Ophthalmol. 2019 Jul;29(4):453-457. doi: 10.1177/1120672118799626. Epub 2018 Sep 11. PMID 30203671